CLINICAL TRIAL: NCT01623583
Title: A Randomized Controlled Study of the Effect of a Needle Phobia or Apprehension Intervention With or Without Synera® on Conversion From Central Venous Catheters to Arteriovenous Fistula or Graft
Brief Title: Effect of Including Synera® in Discussions on Dialysis Access Conversion in Patients With Needle Phobias
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: limited qualifying patient population
Sponsor: Davita Clinical Research (Industry)
Collaborators: Nuvo Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-02-02-NVO-MI
Record Dates: First submitted 2012-05-31; First posted 2012-06-20 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2015-04

CONDITIONS: Needle Phobia; Phobic Disorders
Keywords: lidocaine; tetracaine; Renal dialysis
MeSH Terms: conditions — Phobic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Needle Phobia Intervention (Experimental): Patients will receive enhanced needle phobia intervention comprising the standard intervention plus demonstration of Synera
  Interventions: Other: Enhanced Needle Phobia Intervention
- Standard Needle Phobia Intervention (Active Comparator): Patients will receive the standard intervention for needle phobia
  Interventions: Other: Standard Needle Phobia Intervention

INTERVENTIONS:
Other: Enhanced Needle Phobia Intervention — The enhanced intervention will include the standard intervention, with two enhancements:
  * The video will include a segment with a patient using and discussing the analgesic effects of the Synera patch
  * Before the intervention, a nurse will explain how Synera works and demonstrate its efficacy by having the patient apply it to the non-dominant forearm and leave it in place for 30 minutes, during the intervention. The patient will then be given the opportunity to gently poke 3 times an area of the forearm at least 3 inches from where the patch was applied, and then poke 3 times the center of the area where the patch was applied. The patient may repeat this process up to 3 times. The patient will be asked if he or she can feel the difference in sensitivity.
  Arms: Enhanced Needle Phobia Intervention
Other: Standard Needle Phobia Intervention — The standard intervention will include the following components:
  1. Educational material and discussion with the social worker about the benefits of AVF/AVG over catheter.
  2. Basic training on relaxation breathing
  3. Brief video of a patient overcoming needle phobia
  4. Exposure to a cannulation needle while practicing relaxation breathing, ending in the patients physically holding the needle
  Arms: Standard Needle Phobia Intervention

SUMMARY:
An arteriovenous fistula or graft access (AVF/AVG) for dialysis is often considered a superior option for delivery of dialysis, but requires needles to be inserted. Patients on dialysis who indicate fear of needles as the reason for not switching from a long-term central venous catheter (CVC) access to a fistula or graft access and who otherwise meet the eligibility criterial will be asked to participate. Patients will receive either a standard or an enhanced intervention to address their fear of needles. The enhanced intervention includes the standard intervention plus video training about Synera and trying out an actual patch. Over the 4 months following the intervention, how many patients sign up to switch access will be tracked.

DETAILED DESCRIPTION:
Patients with long-term CVCs (> 180 days) will be recruited for study participation by being asked "Why haven't you gotten a graft or fistula?" Those who indicate fear or discomfort with needles in the top 3 reasons will be consented into the study and administered the AVF/AVG Stages of Change Questionnaire.

The Stages of Change questionnaire has been used extensively in research and has been shown to be highly predictive of people engaging in the behavior of interest. The five stages of change include: 1) Precontemplation: Patient doesn't know about, or knows about but doesn't want to think about, a behavior change; 2) Contemplation: Patients knows about and is beginning to consider behavior change; 3) Planning: Patient is actively investigating and making plans for behavior change; 4) Action: Patient is committed to make the change and/or has taken concrete steps to change behavior; and 5) Maintenance: Patient has made the behavior change and is trying maintain that change.

Patients will be cluster-randomized to receive a standard needle phobia intervention (n = 32), or an enhanced intervention consisting of a standard intervention plus a demonstration of the Synera patch (n = 32) within 15 days of baseline. The intervention will be administered by a study team member. In clinics where there is more than 1 patient randomized to a group, the intervention can be administered to multiple patients simultaneously. The standard intervention will last approximately 20 to 30 minutes. During this time, patients will receive information about the advantages of arteriovenous fistula or graft over central-venous catheter, be taught basic relaxation breathing, see a brief video of a patient overcoming needle fear, and have the opportunity to safely interact with a cannulation needle. In the enhanced intervention, the patient will receive the standard intervention with 2 enhancements: (1) the video will include a segment in which a patient experiences the analgesic effects of the a Synera patch and (2) a Synera patch will be applied at the beginning of the intervention, and 30 minutes later the patient will be given the chance to explore the analgesic effects of Synera.

Patients will complete a Stages of Change questionnaire 1 week after the intervention. Patients will then be followed for 4 months to determine whether or not they have scheduled a vein mapping appointment or have had a fistula or graft access placed.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving hemodialysis at a DaVita clinic/dialysis center
* Receiving in-center hemodialysis thrice weekly
* Central venous catheter (CVC) use for > 180 days
* Patients report a fear of needles as a top-3-reason for failure to get an arteriovenous fistula/graft

Exclusion Criteria:

* Patients have a known intolerance or hypersensitivity to Synera
* Patient with a history of or past diagnosis of severe hepatic disease
* Patient is currently receiving any class 1 antiarrhythmic drugs (i.e., tocainide, mexiletine, etc)
* Patient has a clinically significant illness within 14 days of Screening/Day 1 that, in the opinion of the investigator, would preclude the subject from participating in the study
* Patient has an AVF or AVG in place or is scheduled for placement
* Women and men whose partners are of childbearing potential (defined as premenopausal and not surgically sterilized [ie, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy] or postmenopausal for < 2 years) agree to practice 1 of the following medically acceptable methods of birth control and agree to continue with the regimen throughout the duration of the study: Oral, implantable, or injectable contraceptives for 3 consecutive months before the Screening Visit; Intrauterine device (IUD); and double barrier method (ie, condom, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)
* Patient has significant disease or condition that, in the PI's opinion, may interfere with protocol adherence or subjects' ability to provide informed consent
* Patient is unable to read or comprehend English at a 6th grade level
* Patient has a visual impairment and is unable to read the survey instruments
* Patient has a suspected or known access-related infection at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving a score of 3 or 4 on the stages of change questionnaire | One week after intervention meeting
  The primary outcome measure is how many patients progress from a score of 1 or 2 on the questionnaire (precontemplation or contemplation) as measured before the intervention to a score of 3 or 4 (planning or action) after the intervention, and it is measured one week after the intervention.

SECONDARY OUTCOMES:
Proportion of patients for whom the intervention was successful | Four months after intervention meeting
  The secondary outcome measure will be assessed as a two-stage dichotomous indicator of intervention success. Stage 1 will assess if a patient has had dialysis treatment with a fistula or graft as primary access. If yes, the intervention will be considered a success; if no, stage 2 will ask if the patient has had a vein mapping procedure, which would be considered a success.

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Krishnan, MD, MPH, MBA, Principal Investigator — Davita Clinical Research
Locations (3):
- United States (3):
  - Sunset Dialysis Center, Rancho Cordova, California
  - Natomas Dialysis, Sacramento, California
  - Asheville Kidney Center, Asheville, North Carolina